CLINICAL TRIAL: NCT03949452
Title: Comparative Study Between Subcostal Transversus Abdominis Plane Block Analgesia and Epidural Analgesia in Upper Abdominal Surgeries
Brief Title: Subcostal Transversus Abdominis Plane Versus Epidural Block in Abdominal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD ∕ 17.12.104
Record Dates: First submitted 2019-05-08; First posted 2019-05-14 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2019-05

CONDITIONS: Upper Abdominal Surgery

STUDY DESIGN:
Intervention Model Description: Double blind (participant, investigator) study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcostal Transversus Abdominis Plane catheter (Active Comparator): This group includes patients who will receive subcostal Transversus abdominis plane block analgesia
  Interventions: Other: Subcostal Transversus Abdominis Plane catheter
- Epidural catheter (Placebo Comparator): This group includes patients who will receive epidural analgesia using a catheter technique
  Interventions: Other: Epidural catheter

INTERVENTIONS:
Other: Subcostal Transversus Abdominis Plane catheter — Prior to surgery, an ultrasound guided unilateral Subcostal Transversus abdominis plane bolus dose (consisting of amixture of 10 ml bupivaccaine 0.5% plus 100 mg magnesium sulphate to be completed by normal saline to a total volume of 20 ml mixture) will be given on the same side of the surgical incision.
  At the end of surgery, A Transversus abdominis plane catheter will be inserted unilaterally by surgeon during wound closure. Then postoperatively, Transversus abdominis plane infusion of a solution mixture prepared in multiple 50 cm syringes each syringe contain 20 ml bupivacaine 0.5% plus 100 mg magnesium sulphate to be balanced by normal saline to 50 ml solution mixture ( final concentration of bupivacaine is 0.2%). This solution mixture will be infused through Transversus abdominis plane catheter at a rate of 6 ml/hour for 72 hours postoperatively.
  Arms: Subcostal Transversus Abdominis Plane catheter
Other: Epidural catheter — Prior to surgery, we will site an epidural catheter in the thoracic T7-T9 region, and inject an epidural bolus dose same as described above (consisting of amixture of 10 ml bupivaccaine 0.5% plus 100 mg magnesium sulphate to be completed by normal saline to a total volume of 20 ml mixture) for intra operative analgesia.
  Postoperatively, patients will receive epidural infusion of the solution mixture (same as described above) prepared in multiple 50 cm syringes each syringe contain 20 ml bupivaccaine 0.5% plus 100 mg magnesium sulphate to be balanced by normal saline to 50 ml solution mixture ( final concentration of bupivaccaine is 0.2%). This solution mixture will be infused epidurally at a rate of 6 ml/hour for 72 hours (3 days) postoperatively.
  Arms: Epidural catheter

SUMMARY:
The investegators aimed to compare the efficacy of subcostal Transversus abdominis plane analgesia, to epidural analgesia intra and postoperatively in upper abdominal surgeries.

DETAILED DESCRIPTION:
Epidural analgesia, once considered the gold standard for major abdominal surgeries, but is often associated with sympathetic blockade that creates hypotension and could therefore adversely affect the conduit. Epidural analgesia is recently replaced by other techniques with an improved risk benefit ratio. Pain management techniques that use peripheral nerve blockade are becoming more prevalent, reducing the need for an epidural. Transversus abdominis plane (TAP) approach is aimed to access the nerves in this neurofacial plane between internal oblique muscle and transversus abdominis through the lumbar triangle of Petit. Subcostal Transversus abdominis plane block, has been reported to provide analgesia for incisions extending above the umbilicus. However, there have been few clinical trials on the analgesic efficacy of continuous subcostal Transversus abdominis plane analgesia after major abdominal surgeries. It has been reported recently that supplemental magnesium has a role in providing perioperative analgesia, because this is a relatively harmless molecule, not expensive and because the biological basis for its potential antinociceptive effect is promising. No clinical studies have examined the effect of magnesium sulphate administered continuously in subcostal Transversus abdominis plane catheters as an adjunct to bupivacaine in postoperative analgesia.

The aim of this study is to compare the efficacy of subcostal Transversus abdominis plane analgesia, to epidural analgesia in major upper abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I, II or III
* The incision included is right subcostal incision for major upper abdominal surgeries (partial hepatectomy, pancreatic surgery included Whipple's procedure, total pancreatectomy and distal pancreatectomy) and other operations using the same incision.

Exclusion Criteria:

* Patient refusal.
* Hematological diseases.
* Bleeding diseases.
* Coagulation abnormality.
* Local skin infection
* Sepsis at site of the block.
* Known hypersensitivity to the study drugs.
* Body Mass Index > 35 Kg/m2.
* If the lower end of the incision extended below T10 (umbilicus).
* If the incision extended laterally beyond the anterior axillary line or extended to pass the midline to the other side.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | For 72 hours after surgery
  Intravenous morphine in adose of 0.05 mg/kg will be given if Visual Analogue Scale (VAS) is more than 30 mm in both groups and can be repeated every 15 minutes till Visual Analogue Scale become less than 3. Morphine administration will be ceased when the Visual Analogue Scale score <30 mm on assessment or when over-sedation or respiratory depression occurred (a respiratory rate of < 10 bpm). Doses given will be calculated daily and recorded.

SECONDARY OUTCOMES:
First request for rescue analgesia | for 72 hours after surgery
  First time patient ask for analgesia: in the post anesthesia care unit (PACU) will be recorded and morphine in a dose of 0.05 mg/kg will be given and the time recorded.
Pain Scores | up to 72 hours postoperatively
  * Presence and severity of pain will be assessed in All patients during rest and coughing using visual analogue scale (VAS).
  * Visual analogue scale (VAS) ranging from 0 to 10 while 0 as no pain and 10 as worst imaginable pain.
  * Presence and severity of pain will be assessed at 1, 2, 4, 8, 12, 24, 36, 48, 60 and 72 hours postoperatively.
Heart rate | for 72 hours postoperative
  Heart rate will be assessed at 1, 2, 4, 8, 12, 24, 36, 48, 60 and 72 hours postoperatively.
Mean arterial blood pressure | for 72 hours postoperative
  Mean arterial blood pressure will be assessed at 1, 2, 4, 8, 12, 24, 36, 48, 60 and 72 hours postoperatively.
Peripheral oxygen saturation | for 72 hours postoperative
  Peripheral oxygen saturation will be assessed at 1, 2, 4, 8, 12, 24, 36, 48, 60 and 72 hours postoperatively.
Nausea and vomiting | up to 72 hours postoperatively
  Nausea and vomiting: will be assessed through nausea scores (none = 0, mild = 1, moderate = 2 and vomiting = 3) at 1, 2, 4, 8, 12, 24, 36, 48, 60,72 hrs post operativly. We offered rescue antiemetics to any patient who had a nausea score of 2 or more.
Degree of sedation | for 72 hours postoperative
  Degree of sedation will be assessed by using the sedation scale described by Culebras (2001) as:
  * 1 : Awake and alert,
  * 2 : Sedated, responding to verbal stimulus,
  * 3 : Sedated, responding to mild physical stimulus,
  * 4 : Sedated, responding only to moderate or severe physical stimulus
  Degree of sedation will be assessed at 1, 2, 4, 8, 12, 24, 36, 48, 60 and 72 hours postoperatively
Serum level of magnesium sulphate | up to 72 hours postoperatively
  Degree of sedation will be assessed by using the sedation scale described by Culebras (2001) as:
  * 1 : Awake and alert,
  * 2 : Sedated, responding to verbal stimulus,
  * 3 : Sedated, responding to mild physical stimulus,
  * 4 : Sedated, responding only to moderate or severe physical stimulus
  Degree of sedation will be assessed at 1, 2, 4, 8, 12, 24, 36, 48, 60 and 72 hours postoperatively
Patient satisfaction with their analgesia | up to 72 hours postoperatively
  * Patient satisfaction with their analgesia will be assessed as (poor = 1, fair = 2, good = 3, excellent = 4).
  * Patient satisfaction with their analgesia will be assessed at 24, 48 and 72 hours post operatively.
Wound pain | up to 3 months postoperatively
  * Residual or chronic wound pain will be assessed in All patients using visual analogue scale (VAS).
  * Visual analogue scale (VAS) ranging from 0 to 10 while 0 as no pain and 10 as worst imaginable pain.
  * Residual wound pain will be assessed at 30, 60, 90 days postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Y Makharita, MD, Study Chair — Professor of Anesthesia and Surgical Intensive Care; Hazem ES Moawad, MD, Study Director — Assistant Professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol
Time Frame: data will be available within 6 monthes of study completion.
Access Criteria: Data may be shared by contacting the principle investegator.

REFERENCES:
- [Result] Hebbard P. Subcostal transversus abdominis plane block under ultrasound guidance. Anesth Analg. 2008 Feb;106(2):674-5; author reply 675. doi: 10.1213/ane.0b013e318161a88f. No abstract available. PMID 18227342
- [Result] Culebras X, Van Gessel E, Hoffmeyer P, Gamulin Z. Clonidine combined with a long acting local anesthetic does not prolong postoperative analgesia after brachial plexus block but does induce hemodynamic changes. Anesth Analg. 2001 Jan;92(1):199-204. doi: 10.1097/00000539-200101000-00038. PMID 11133627